CLINICAL TRIAL: NCT03814161
Title: FRailty Among Elderly Emergency Department Patients With Outcome Measures
Acronym: FREEDOM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: FREEDOM
Record Dates: First submitted 2018-10-12; First posted 2019-01-23 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Geriatric, Frailty, Emergency Department
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to compare 4 clinical frailty scores, namely Clinical Frailty Scale (CFS), Edmonton Frail Scale (EFS), FRAIL 5-item scale (FRAIL) and SARC-F Sarcopenia Score (SARC-F), which can potentially be adopted for daily practice in the busy ED. It is timely as we projected that we will be seeing more elderly patients attending the ED for various medical and surgical conditions. Their attendance at the ED would be a good opportunity to screen for frailty among them, and to intervene to prevent adverse outcomes such as ED re-attendance or subsequent hospitalisation that might lead to poor functional outcomes and higher dependence on step-down care facilities.

ELIGIBILITY:
Inclusion Criteria:

- Elderly patients aged 65 years and above attending ED irrespective of reason for attendance.

Exclusion Criteria:

* Haemodynamically unstable patients
* Inability to obtain informed consent
* Inability to obtain reliable information from patient or caregiver (e.g. deafness, blindness, language barriers)
* Vulnerable populations (e.g. prisoners)
* Patients who are planned for hospital admission from the ED

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 years and above attending Emergency Department, National University Hospital, Singapore irrespective of reason for attendance and are planned for discharge from the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
1-month Adverse Event Occurrence (composite) | At 1 month after index ED visit
  Falls, ED re-attendance, hospital/ nursing home admission, decline in Activities of Daily Living and/or all-cause mortality

SECONDARY OUTCOMES:
3-month Adverse Event Occurrence (composite) | At 3 months after index ED visit
  Falls, ED re-attendance, hospital/ nursing home admission, decline in Activities of Daily Living and/or all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wei Yau, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209